CLINICAL TRIAL: NCT02886988
Title: A Randomized, Placebo-Controlled, Double-Blind, Prospective Clinical Trial of Botulinum Toxin Type A in Prevention of Hypertrophic Scar Development in Median Sternotomy Wound
Brief Title: Early Postoperative Prevention and Treatment of Median Sternotomy Scars With Botulinum Toxin Type A Injection
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KY20162057-2
Record Dates: First submitted 2016-08-29; First posted 2016-09-01 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2016-08

CONDITIONS: Scar
Keywords: Botulinum toxin type A, scar
MeSH Terms: conditions — Cicatrix | interventions — Botulinum Toxins, Type A; Botulinum Toxins; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Botulinum toxin type A (Experimental): The entire median sternotomy wound was divided into the upper half and the lower half. Both halves of the wound were randomized to receive treatment with either BTA or 0.9% normal saline.100U Botulinum toxin type A(BTA) will be reconstituted with 2mL of normal saline for a concentration of 50U/mL. 0.1ml(5 units) of BTA will be injected along the wound edges. The injections will be administered within 14 days of median sternotomy with a 30G needle.
  Interventions: Drug: Botulinum toxin type A
- Normal Saline (Placebo Comparator): The entire median sternotomy wound was divided into the upper half and the lower half. Both halves of the wound were randomized to receive treatment with either BTA or 0.9% normal saline.0.1ml normal saline will be injected along the wound edges.
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Botulinum toxin type A — 50 units of botulinum toxin diluted in 1 ml of normal saline will be administered. 0.1mlof BTA will be injected with a 30G needle.
  Other Names: Botox; Botulinum Toxin
  Arms: Botulinum toxin type A
Drug: normal saline — 0.1mlof normal saline will be injected with a 30G needle.
  Other Names: NaCl 0.9%
  Arms: Normal Saline

SUMMARY:
Linear hypertrophic scar is a common surgical problem that can be difficult to manage, especially for the median sternotomy scar. Despite high demand for the early intervention to prevent and treat surgical scars, there is yet no universal consensus on satisfactory treatment. Botulinum toxin type A is a neurotoxin that has been widely and safely used in medicine for more than 30 years. It induces chemodenervation through acting on the presynaptic neuron to prevent release of acetylcholine, which leads to functional denervation of striated muscle for about 6 months after injection. The aim of this randomized controlled trial is to evaluate the efficacy of Botulinum toxin type A as a prophylactic treatment in the early postoperative of median sternotomy for the purpose of preventing excess scar formation.

DETAILED DESCRIPTION:
The goal of this study is to conduct a randomized controlled trial about using Botulinum toxin type A ( BTA) to prevent hypertrophic scar in median sternotomy wound. The entire median sternotomy wound was divided into the upper half and the lower half. Both halves of the wound were randomized to receive treatment with either BTA or 0.9% normal saline. The patient and the surgeon will be blinded to the treatment arm. The primary end point was the evaluation of upper and lower half scar using the Vancouver Scar Scale (VSS). At 6 months follow-up, two blinded dermatologists examined the patients and took photographs of the scar in the outpatient clinic of XiJing Hospital. Scars were assessed using the VSS and assigned the mean score of the two observers. At 6-month follow-up, ultrasonography to measure the scar width will be performed. At the same time, patients were asked to evaluate their overall satisfaction, using a four-point grading scale for each half the scar(1= very satisfied, 2= satisfied,3= slightly satisfied, 4= unsatisfied ).Paired t-test was used to compare the VSS scores, scar width and the overall satisfaction between the BTA-treated group and normal saline group.

ELIGIBILITY:
Inclusion Criteria:

* Patients included are older than 18 years with a median sternotomy less than 14 days.
* Patients are willing and able to participate in the study as an outpatient, making several visits to the study center during the treatment and follow-up periods.
* Patients can comply with all study requirements including concomitant medication and other treatment restrictions.
* Patients have good wound healing condition, without infection sign.

Exclusion Criteria:

* The exclusion criteria applied is current pregnancy or breast feeding, allergy to botulinum toxin type A, previous injection of botulinum toxin within 6 months prior to enrollment, Myasthenia gravis or other neuromuscular disorder,and refusal to participate in this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-10; Primary Completion 2017-12-28 (Actual); Study Completion 2018-01-22 (Actual)

PRIMARY OUTCOMES:
Vancouver scar scale | 6 months after Botulinum toxin type A injection
  Vancouver scar scale measures pigmentation, vascularity, pliability and scar height 6 months after received BTA injection.

SECONDARY OUTCOMES:
Scar width | 6 months after Botulinum toxin type A injection
  At 6-month follow-up, scar width will be measured by ultrasonography.
Patient satisfaction | 6 months after Botulinum toxin type A injection
  At 6-month follow-up, patients were asked to evaluate their overall satisfaction, using a four-point grading scale for each half the scar.

CONTACTS AND LOCATIONS:
Overall Officials: Song-Tao Xie, Principal Investigator — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ozog DM, Moy RL. Discussing Fractional Carbon Dioxide Laser and Other Physical Treatments for Scar Prevention With Patients. JAMA Dermatol. 2015 Aug;151(8):815-6. doi: 10.1001/jamadermatol.2015.0594. No abstract available. PMID 25946625
- [Background] Kim YS, Lee HJ, Cho SH, Lee JD, Kim HS. Early postoperative treatment of thyroidectomy scars using botulinum toxin: a split-scar, double-blind randomized controlled trial. Wound Repair Regen. 2014 Sep-Oct;22(5):605-12. doi: 10.1111/wrr.12204. Epub 2014 Aug 26. PMID 24898579
- [Background] Zhang DZ, Liu XY, Xiao WL, Xu YX. Botulinum Toxin Type A and the Prevention of Hypertrophic Scars on the Maxillofacial Area and Neck: A Meta-Analysis of Randomized Controlled Trials. PLoS One. 2016 Mar 17;11(3):e0151627. doi: 10.1371/journal.pone.0151627. eCollection 2016. PMID 26985661
- [Background] Elhefnawy AM. Assessment of intralesional injection of botulinum toxin type A injection for hypertrophic scars. Indian J Dermatol Venereol Leprol. 2016 May-Jun;82(3):279-83. doi: 10.4103/0378-6323.173586. PMID 27088929
- [Background] Shaarawy E, Hegazy RA, Abdel Hay RM. Intralesional botulinum toxin type A equally effective and better tolerated than intralesional steroid in the treatment of keloids: a randomized controlled trial. J Cosmet Dermatol. 2015 Jun;14(2):161-6. doi: 10.1111/jocd.12134. Epub 2015 Mar 24. PMID 25810045
- [Background] Prodromidou A, Frountzas M, Vlachos DE, Vlachos GD, Bakoyiannis I, Perrea D, Pergialiotis V. Botulinum toxin for the prevention and healing of wound scars: A systematic review of the literature. Plast Surg (Oakv). 2015 Winter;23(4):260-4. doi: 10.4172/plastic-surgery.1000934. PMID 26665143
- [Background] Jeong HS, Lee BH, Sung HM, Park SY, Ahn DK, Jung MS, Suh IS. Effect of Botulinum Toxin Type A on Differentiation of Fibroblasts Derived from Scar Tissue. Plast Reconstr Surg. 2015 Aug;136(2):171e-178e. doi: 10.1097/PRS.0000000000001438. PMID 26218391
- [Background] Chen M, Yan T, Ma K, Lai L, Liu C, Liang L, Fu X. Botulinum Toxin Type A Inhibits alpha-Smooth Muscle Actin and Myosin II Expression in Fibroblasts Derived From Scar Contracture. Ann Plast Surg. 2016 Sep;77(3):e46-9. doi: 10.1097/SAP.0000000000000268. PMID 25144422